CLINICAL TRIAL: NCT02643394
Title: The Comparative Efficacy of Oral vs. Intravenous Acetaminophen in Sinus Surgery Patients
Brief Title: Efficacy of Oral vs. Intravenous Acetaminophen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 052015-068
Record Dates: First submitted 2015-06-02; First posted 2015-12-31 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain
Keywords: Acetaminophen; Postoperative pain; Sinus Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Acetaminophen (Active Comparator): Oral Acetaminophen 1-hour before surgery
  Interventions: Drug: Oral Acetaminophen
- Intravenous Acetaminophen (Active Comparator): Intravenous Acetaminophen within 1-hour prior to anesthetic emergence
  Interventions: Drug: Intravenous acetaminophen

INTERVENTIONS:
Drug: Oral Acetaminophen — 1000mg oral acetaminophen + 400mg oral celecoxib given within one hour of incision
  Other Names: Tylenol
  Arms: Oral Acetaminophen
Drug: Intravenous acetaminophen — 400mg oral celecoxib given within one hour of incision + 1000mg IV acetaminophen within one hour prior to anesthetic emergence.
  Other Names: Tylenol
  Arms: Intravenous Acetaminophen

SUMMARY:
The comparative efficacy of intravenous (IV) to oral (PO-'per os') acetaminophen in the management of postoperative pain is understudied and largely unknown. In this observer blinded randomized clinical trial, investigators aim to determine the comparative efficacy of PO (preoperative) vs. IV (intraoperative) acetaminophen in a sinus surgery population.

DETAILED DESCRIPTION:
The comparative efficacy of intravenous (IV) to oral (PO-'per os') acetaminophen is understudied and largely unknown. Intravenous acetaminophen has been available since 2010 (http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/022450lbl.pdf) and has proven superiority over placebo in human clinical trials. It is clearly advantageous in patients who cannot take oral medications. Similarly, oral acetaminophen has proven efficacy in the management of postoperative pain.

However, in patients who can receive either formulation the incremental cost of the IV formulation, both to the Health System and patient, is substantial. This incremental cost would be justifiable if there were clear efficacy or safety data to support the preferential use of IV over PO acetaminophen.

However, there is no evidence of superior safety and there are only two studies to our knowledge investigating the question of comparative efficacy. Fenlon et al. randomized 130 patients undergoing 3rd molar (i.e., wisdom tooth) removal to IV vs. PO acetaminophen and found that PO acetaminophen was non-inferior to IV acetaminophen. The primary endpoint was postoperative pain score 1h after surgery. No safety concerns were identified in either group. Pettersson et al. randomized cardiac surgery patients to IV or PO acetaminophen, starting immediately postoperatively through the following morning, and found a significant opioid sparing effect of IV acetaminophen but no difference in pain scores or nausea.

IV acetaminophen avoids first-pass hepatic metabolism and therefore generates higher serum and cerebrospinal fluid (CSF)/brain levels than does PO acetaminophen (http://ofirmev.com/Pharmacokinetics/). Based on the pharmacokinetic data, one can hypothesize that IV acetaminophen would be superior to PO acetaminophen at time points where serum and/or cerebrospinal fluid drug levels are higher.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Undergoing elective sinus surgery at Zale Lipshy Hospital

Exclusion Criteria:

* Inability of the patient to follow directions or comprehend either English or Spanish language.

  * Disorders of the liver which would make acetaminophen contraindicated (such as hepatitis, liver failure, prior liver transplant, etc).
  * Patients with chronic pain manifest by a baseline pain score > 4/10
  * Chronic opioid use (>2 weeks continuously), or illicit drug abuse
  * Body weight < 50 kg.
  * Patients with contraindications to any of the study drugs (such as Malignant Hyperthermia susceptible, celecoxib or sulfa allergy, etc.).
  * Patients who have taken analgesic medications on the morning of surgery (prior to arrival).
  * Allergy to acetaminophen

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2018-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David McDonagh, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Zale Lipshy University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Started | 55 | 55
Completed | 51 | 50
Not Completed | 4 | 5
Not completed — Protocol Violation | 4 | 5

BASELINE CHARACTERISTICS:
Population: Adult patients undergoing sinus surgery at a single major academic medical center
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 42 | 86
  >=65 years | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (16.3) | 54.0 (15.7) | 52.7 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 34 | 35 | 69
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score on the Scale of 10 (0=No Pain and 10=Worst Pain)
Description: Pain score on the scale of 10 at 1-h postoperatively in the Post-Anesthesia Care Unit (PACU)
Time Frame: 1-h postoperatively
Population: Subjects undergoing Functional Endoscopic Sinus Surgery were enrolled to the study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 51 | 50
units on a scale | 2 [0 to 3] | 2 [0 to 5]
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.252, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Morphine Equivalents of Postoperative Opioid Usage
Description: Total amount of postoperative opioid usage at Postoperative Anesthesia Care Unit (PACU), an expected average of 6 hours
Time Frame: an expected average of 6 hours
Population: Subjects undergoing Functional Endoscopic Sinus Surgery were enrolled to the study.
Measure: Median (Inter-Quartile Range); unit: Morphine equivalent (mg)
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 51 | 50
Morphine equivalent (mg) | 5 [0 to 10] | 5 [0 to 14.8]
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.402, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Through 24h post-operatively
Description: Patient phone call at 24h
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/50
Other Adverse Events (participants affected / at risk) | 3/51 | 6/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Acetaminophen (N=51) | Intravenous Acetaminophen (N=50)
Nausea (Gastrointestinal disorders) | 3 (3) | 6 (6) — Nausea following PACU discharge (assessed at 24h post-operatively)

LIMITATIONS AND CAVEATS:
Single center Sinus surgery population only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes